CLINICAL TRIAL: NCT03097848
Title: Efficacy and Safety of Combination of Sorafenib as Preoperative Adjuvant and Latter Radiofrequency Ablation in the Treatment Of Recurrent Hepatocellular Carcinoma: A Prospective Multicenter Cohort Study
Brief Title: Efficacy and Safety of Sorafenib as Adjuvant and Latter Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma
Acronym: ESCALATOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Chengdu PLA General Hospital (Other); Sichuan Provincial People's Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Hunan Cancer Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); The First People's Hospital of Yunnan (Other); Yunnan Cancer Hospital (Other); Xiangya Hospital of Central South University (Other); Xinqiao Hospital of Chongqing (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Henan Cancer Hospital (Other Government); First Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, feng xiaobin, Clinical Professor, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWHB 019
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: HCC
MeSH Terms: interventions — Control Groups; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib+RFA group (Experimental): for eligible cases, combination treatment with RFA and Sorafenib will be given.That is sorafenib for 2 week,then radiofrequency ablation
  Interventions: Procedure: RFA; Drug: Sorafenib
- RFA group (Active Comparator): for eligible cases, RFA will be given only.
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — for eligible cases, radiofrequency ablation will be given only.
  Other Names: control group
Drug: Sorafenib — for eligible cases, combination treatment with RFA and Sorafenib will be given.That is sorafenib for 2 week,then radiofrequency ablation
  Other Names: experimental group
  Arms: Sorafenib+RFA group

SUMMARY:
Radiofrequency ablation is a popular treatment for recurrent hepatocellular carcinoma (HCC),but still has a higher recurrence. Sorafenib as neo-adjuvant therapy in combination of RFA was not reported yet. There's a theoretical advantage of this combination. Hence in this study the efficacy and safety of pre-administrative Sorafenib and Latter radiofrequency ablation (RFA) in Recurrent HCC will be tested in a multicenter prospective cohort study.

DETAILED DESCRIPTION:
Radiofrequency ablation is a popular treatment for recurrent hepatocellular carcinoma (HCC),but still has a higher recurrence. Sorafenib as neo-adjuvant therapy in combination of RFA was not reported yet. There's a theoretical advantage of this combination. Hence in this study the efficacy and safety of pre-administrative Sorafenib and Latter radiofrequency ablation (RFA) in Recurrent HCC will be tested in a multicenter prospective cohort study. Eligible cases will be assigned into the experimental group and the control group. For experiment group, sorafenib tablet will be given for two weeks, and then perform radiofrequency ablation. For the control group, RFA will be performed immediately.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 75 years old
* Without gender restriction
* With a favorable liver function of Child-Pugh A to B
* No contraindications to RFA and anesthesia
* Diagnosed with Recurrent HCC
* Signed informed consent.

Exclusion Criteria:

* Cancer thrombosis in major vessels/ extrahepatic metastasis
* Uncontrollable ascites or variceal bleeding
* Impairment in liver function
* Severe disorders in vital organ
* Accompanied with other tumors or infectious disease except hepatitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 1 year
  1 year Disease free survival

SECONDARY OUTCOMES:
Time To Recurrence | 3 year
  time to tumor recurrence
Overall Survival | 3 year
  overall survival
postoperative complications | 6 months
  postoperative complications diagnosed within 6 months
Health economics index | 3 years
  Health economics index within 3 years
mortality | 3 months
  mortality occured within 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided